CLINICAL TRIAL: NCT00960986
Title: A Phase 4 Comparison of Duloxetine Dosing Strategies in the Treatment of Korean Patients With Major Depressive Disorder
Brief Title: A Duloxetine Dosing Strategy Study in Korean Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9884; F1J-MC-HMFL (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2012-04-17 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Duloxetine 60 mg with food (Experimental): Duloxetine 60 milligram (mg) capsule oral (po), once daily (QD) with food for 8 weeks
  Interventions: Drug: Duloxetine hydrochloride
- Duloxetine 60 mg without food (Experimental): Duloxetine 60 mg capsule po QD without food for 8 weeks
  Interventions: Drug: Duloxetine hydrochloride
- Duloxetine 30 mg with food (Experimental): Duloxetine 30 mg capsule po QD with food for 1 week, then 60 mg with food for 7 weeks
  Interventions: Drug: Duloxetine hydrochloride
- Duloxetine 30 mg without food (Experimental): Duloxetine 30 mg capsule po QD without food for 1 week, then 60 mg without food for 7 weeks
  Interventions: Drug: Duloxetine hydrochloride

INTERVENTIONS:
Drug: Duloxetine hydrochloride — po, QD
  Other Names: Cymbalta; LY248686

SUMMARY:
The purpose of this study is to assess nausea severity in response to four different drug dosing strategies of Duloxetine (30 mg with food, 60 mg with food, 30 mg without food, and 60 mg without food) in Korean patients with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* For females of child-bearing potential test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.
* 17-item Hamilton Depression Rating Scale (HAMD-17) total score >15 at Screening and Randomization
* Have signed the informed consent document (ICD)
* Have a level of understanding sufficient to provide informed consent and to communicate with the investigators and site personnel
* Are judged to be reliable and agree to keep all appointments for clinic visits, tests, and procedures required by the protocol
* Patients must meet Diagnostic and Statistical Manual of Mental Disorders-fourth edition-text revision (DSM-IV-TR) criteria for Major Depressive Disorder (MDD). The Mini International Neuropsychiatric Interview (MINI) will be used to establish the diagnosis and exclude other psychiatric illnesses.

Exclusion Criteria:

* Treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have any current primary Axis I disorder other than MDD
* Have any previous diagnosis of bipolar disorder, schizophrenia, or other psychotic disorders
* Lack of response of the current episode of major depression to two or more adequate courses of antidepressant therapy at clinically appropriate dose for a minimum of 4 weeks or, in the judgment of the investigator, the patient meets criteria for treatment-resistant depression
* Have a history of a lack of response, at any time, to an adequate trial of duloxetine (defined as treatment with at least 60 mg/day of duloxetine for a minimum of 4 weeks)
* Presence of an Axis II disorder that, in the judgment of the investigator, would interfere with study compliance
* DSM-IV-TR-defined history of substance abuse or dependence within the past 6 months, excluding nicotine and caffeine
* Patients judged to be at serious suicidal risk in the opinion of the investigator and/or score ≥3 on Item 3 (suicide) of the HAMD-17
* Serious medical illness or clinically significant laboratory abnormalities that, in the judgment of the investigator, are likely to require intervention/hospitalization/excluded medication during the course of the study Note: Patients with acute liver injury (such as hepatitis) or severe (Child-Pugh Class C) cirrhosis will be excluded
* Have an acute or chronic medical illness with the main symptoms of nausea or gastrointestinal discomfort or taking any medication known to have major gastric effects that would interfere with nausea ratings.
* Electroconvulsive therapy (ECT) or Transcranial Magnetic Stimulation (TMS) within the past year
* Taking any excluded medications within 7 days prior to Randomization.
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to Randomization or potential need to use a MAOI within 5 days after discontinuation of study drug.
* Treatment with fluoxetine within 30 days prior to Randomization.
* Frequent and/or severe allergic reactions with multiple medications or known hypersensitivity to duloxetine.
* Abnormal thyroid stimulating hormone (TSH) concentration. Note: Participants diagnosed with hyperthyroidism or hypothyroidism who were treated with a stable dose of thyroid supplement for at least the past 3 months, have medically appropriate TSH concentration, and are clinically euthyroid, are allowed to enroll in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time (UTC/GMT - 5hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- South Korea (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheong Ju-City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goyang-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seongnam-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sungnam-Si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yangsan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period 1 was a 3- to 30-day screening and washout period; Period 2 (Week 0-1) was a 1-week initial dosing period (randomization to duloxetine 30 mg with food, 30 mg without food, 60 mg with food, or 60 mg without food); Period 3 (Week 1-8) was a 7-week therapy period (treatment switched to duloxetine 60 mg once daily (QD) until study end.
Period: Period 1 (Screening and Washout)
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Started | 59 | 63 | 63 | 64
Completed | 56 | 59 | 59 | 61
Not Completed | 3 | 4 | 4 | 3
Not completed — Adverse Event | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 1
Period: Period 2 (1-week Initial Dosing Period)
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Started | 56 | 59 | 59 | 61
Completed | 56 | 59 | 59 | 61
Not Completed | 0 | 0 | 0 | 0
Period: Period 3 (7-week Therapy Period)
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Started | 56 | 59 | 59 | 61
Completed | 26 | 36 | 39 | 36
Not Completed | 30 | 23 | 20 | 25
Not completed — Adverse Event | 17 | 15 | 10 | 12
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 10 | 4 | 3 | 11
Not completed — Withdrawal by Subject | 2 | 2 | 4 | 2
Not completed — Lack of Efficacy | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food | Total
Number analyzed (Participants) | 59 | 63 | 63 | 64 | 249
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 44.65 [31.58 to 53.73] | 47.90 [38.65 to 58.90] | 49.94 [40.04 to 62.24] | 44.65 [32.84 to 56.92] | 46.81 [34.78 to 59.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 47 | 47 | 40 | 177
  Male | 16 | 16 | 16 | 24 | 72
Race/Ethnicity, Customized [Number; unit: participants]
  Korean | 59 | 63 | 63 | 64 | 249
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 59 | 63 | 63 | 64 | 249
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] — BMI measures the participant's body weight divided by the square of his or her height.
  kilogram per square meter (kg/m^2) | 24.56 (4.034) | 23.28 (3.133) | 23.06 (3.430) | 23.84 (3.612) | 23.67 (3.584)
Previously diagnosed with major depressive disorder (MDD) [Number; unit: participants] | 59 | 63 | 63 | 64 | 249
Duration since first major depressive disorder (MDD) episode [Median (Inter-Quartile Range); unit: years] | 1.47 [0.52 to 4.29] | 2.65 [0.77 to 5.32] | 2.52 [0.48 to 9.12] | 1.29 [0.52 to 4.40] | 1.92 [0.54 to 5.55]
Age at first major depressive disorder (MDD) episode [Mean (Inter-Quartile Range); unit: years] | 41.21 [29.00 to 51.00] | 43.33 [34.67 to 53.00] | 43.86 [27.00 to 59.60] | 41.58 [29.00 to 54.00] | 42.52 [30.00 to 54.00]
Number of previous MDD episodes/exacerbations in the last 24 months [Median (Inter-Quartile Range); unit: number of episodes in last 24 months] | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0]
Received previous therapy for current episode [Number; unit: participants]
  yes | 18 | 25 | 18 | 26 | 87
  no | 41 | 38 | 45 | 38 | 162
17-item Hamilton Depression Rating Scale (HAMD-17) Total Score [Mean (Standard Deviation); unit: units on a scale] — The HAMD-17 measured depression severity. Each item was evaluated and scored using either a 5-point scale (for example, absent; mild; moderate; severe; very severe) or a 3-point scale (for example, absent; mild; marked). The total score ranged from 0 (not at all depressed)-52 (severely depressed).
  units on a scale | 21.0 (5.18) | 22.3 (5.69) | 22.9 (5.45) | 20.3 (5.23) | 21.6 (5.46)
Clinical Global Impression of Severity (CGI-S) Score [Mean (Inter-Quartile Range); unit: units on a scale] — The CGI-S Rating Scale was a 7-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill.
  units on a scale | 4.4 [4.0 to 5.0] | 4.5 [4.0 to 5.0] | 4.7 [4.0 to 5.0] | 4.2 [4.0 to 5.0] | 4.4 [4.0 to 5.0]
Association for Methodology and Documentation in Psychiatry (AMDP-5) Item 112 (Nausea) Score [Mean (Standard Deviation); unit: units on a scale] — AMDP-5 Item 112 (nausea) measured nausea severity. The scores ranged from 0-3: 0=Not present; 1=Mild; 2=Moderate; 3=Severe.
  units on a scale | 0.3 (0.72) [0.0 to 0.0] | 0.2 (0.59) [0.0 to 0.0] | 0.2 (0.61) [0.0 to 0.0] | 0.1 (0.38) [0.0 to 0.0] | 0.2 (0.58) [0.0 to 0.0]

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Nausea Severity, Association for Methodology and Documentation in Psychiatry (AMDP-5) Adverse Event (AE) Scale Item 112 (Nausea)
Description: AMDP-5 AE scale Item 112 (nausea) measured nausea severity during treatment (Week 0-8). The scores ranged from 0-3: 0=Not present; 1=Mild; 2=Moderate; 3=Severe.
Time Frame: 1 week and 8 weeks
Population: The safety population included all participants who took at least 1 study drug dose analysed according to the drug dose actually taken.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  Week 0-1 | 1.4 [1.06 to 1.69] | 1.2 [0.89 to 1.49] | 0.9 [0.62 to 1.11] | 0.8 [0.57 to 1.06]
  Week 1-8 (n=35; n=43; n=48; n=46) | 0.5 [0.25 to 0.67] | 0.5 [0.27 to 0.66] | 0.7 [0.45 to 0.96] | 0.4 [0.19 to 0.59]

2. Secondary Outcome: Mean Change From Baseline to 8-Week Endpoint in Association for Methodology and Documentation in Psychiatry (AMDP-5) Adverse Event (AE) Scale Item 112 (Nausea)
Description: Scores for AE scale Item 112 (nausea) of AMDP-5 (Week 0-8) ranged from 0-3: 0=Not present; 1=Mild; 2=Moderate; 3=Severe. Least Squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariate matrix.
Time Frame: Baseline, 8 weeks
Population: The safety population included all participants who took at least 1 study drug dose analysed according to the drug dose actually taken. N = number of subjects with a baseline and post-baseline result at the Week 8 visit.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 28 | 37 | 39 | 37
units on a scale | -0.02 (0.08) | -0.02 (0.07) | -0.01 (0.07) | -1.12 (0.07)

3. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in Association for Methodology and Documentation in Psychiatry (AMDP-5) Measure: Gastric Events Score
Description: Gastric events scores (average of Item 112 [nausea] + Item 113 [vomiting]) of AMDP-5 (Week 0-8) ranged from 0-3: 0=Not present; 1=Mild; 2=Moderate; 3=Severe. Least Squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariate matrix.
Time Frame: Baseline, 1 week and 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | 0.73 (0.10) | 0.72 (0.10) | 0.35 (0.10) | 0.37 (0.10)
  8-week change (n=28; n=37; n=39; n=37) | -0.04 (0.04) | -0.04 (0.04) | -0.04 (0.04) | -0.09 (0.04)

4. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in Association for Methodology and Documentation in Psychiatry (AMDP-5) Measure: Common Adverse Events (AEs) Score
Description: AMDP-5 common AEs score was used to create a composite measure of AEs from previous duloxetine studies (incidence >5% and 2X placebo rate). The common AEs total score was the sum of the following 8 AMDP-5 items: 1) Mean of Item 112 (nausea) + 113 (vomiting); 2) Item 111 (dry mouth); 3) Item 115 (constipation); 4) Mean of Items 101-104 (insomnia); Item 122 (increased perspiration); 8) Item 106 (decreased appetite). Score was based on a 5-point scale: 1=absent, 2=mild, 3=moderate, 4=severe, 5=extremely severe; Higher score=worse severity.
Time Frame: Baseline, 1 week, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | 1.25 (0.44) | 1.28 (0.42) | -0.00 (0.43) | -0.37 (0.41)
  8-week change (n=28; n=37; n=39; n=37) | -3.54 (0.47) | -2.99 (0.42) | -2.33 (0.41) | -3.23 (0.41)

5. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in 17-Item Hamilton Depression Rating Scale (HAMD-17) Total Score
Description: The HAMD-17 total score ranged from 0 (not at all depressed)-52 (severely depressed). Least squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariance matrix.
Time Frame: Baseline, 1 week, 8 weeks
Population: The efficacy population included the number of participants with baseline and at least 1 post-baseline value analysed under the intent-to-treat (ITT) principle according to the drug dose they were assigned.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | -2.83 (0.57) | -2.85 (0.55) | -3.84 (0.56) | -4.34 (0.54)
  8-week change (n=28; n=37; n=39; n=37) | -15.39 (1.01) | -13.45 (0.90) | -13.60 (0.88) | -13.07 (0.89)

6. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in 17-Item Hamilton Depression Rating Scale (HAMD-17) Maier Subscale
Description: The HAMD-17 Maier subscale (Items 1, 2, 7, 8, 9, 10 of HAMD-17 questionnaire) represented the "core" symptoms of depression. Total subscale scores ranged from 0 (normal)-24 (severe). Least Squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariate matrix.
Time Frame: Baseline, 1 week, 8 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | -2.06 (0.33) | -1.90 (0.32) | -2.15 (0.32) | -2.64 (0.31)
  8-week change (n=28; n=37; n=39; n=37) | -8.01 (0.50) | -7.12 (0.45) | -7.55 (0.44) | -7.30 (0.44)

7. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in 17-Item Hamilton Depression Rating Scale (HAMD-17) Core Mood Subscale
Description: The HAMD-17 Core Mood subscale (Items 1, 2, 3, 7, 8 of HAMD-17 questionnaire) represented the core symptoms of depression. Total subscale scores ranged from 0 (normal)-20 (severe). Least Squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariate matrix.
Time Frame: Baseline, 1 week, 8 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | -1.43 (0.27) | -1.18 (0.26) | -1.52 (0.26) | -1.76 (0.25)
  8-week change (n=28; n=37; n=39; n=37) | -6.18 (0.40) | -5.39 (0.36) | -5.85 (0.35) | -5.67 (0.35)

8. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in 17-Item Hamilton Depression Rating Scale (HAMD-17) Anxiety/Somatization Subscale
Description: The HAMD-17 Anxiety/Somatization subscale (Items 10, 11, 12, 13, 15, 17 of HAMD-17 questionnaire) evaluated the severity of psychic and somatic manifestations of anxiety and agitation. Total subscale scores ranged from 0 (normal)-18 (severe). Least Squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariate matrix.
Time Frame: Baseline, 1 week, 8 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | -0.75 (0.25) | -1.15 (0.24) | -1.36 (0.24) | -1.41 (0.23)
  8-week change (n=28; n=37; n=39; n=37) | -4.93 (0.41) | -4.50 (0.36) | -4.57 (0.35) | -4.26 (0.35)

9. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in 17-Item Hamilton Depression Rating Scale (HAMD-17) Retardation/Somatization Subscale
Description: The HAMD-17 Retardation/Somatization subscale (Items 1, 7, 8, 14 of HAMD-17 questionnaire) evaluated dysfunction in mood, work, sexual activity, and overall motor retardation. Total subscale scores ranged from 0 (normal)-14 (severe). Least Squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariate matrix.
Time Frame: Baseline, 1 week, 8 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | -0.83 (0.22) | -0.87 (0.21) | -1.02 (0.22) | -1.20 (0.21)
  8-week change (n=28; n=37; n=39; n=37) | -4.92 (0.35) | -4.37 (0.31) | -4.63 (0.31) | -4.55 (0.31)

10. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in 17-Item Hamilton Depression Rating Scale (HAMD-17) Sleep Subscale
Description: The HAMD-17 Sleep subscale (Items 4, 5, 6 of HAMD-17 questionnaire) evaluated initial, middle, and late insomnia. Total subscale scores ranged from 0 (no difficulty)-6 (difficulty). Least Squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariate matrix.
Time Frame: Baseline, 1 week, 8 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | -0.72 (0.21) | -0.64 (0.21) | -0.66 (0.21) | -1.01 (0.20)
  8-week change (n=28; n=37; n=39; n=37) | -2.77 (0.27) | -2.32 (0.24) | -2.09 (0.23) | -2.10 (0.23)

11. Secondary Outcome: Mean Change From Baseline to 1-Week and 8-Week Endpoints in Clinical Global Impressions of Severity (CGI-S)
Description: The CGI-S Rating Scale was a 7-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; or 7=extremely ill. Least squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction, and an unstructured covariance matrix.
Time Frame: Baseline, 1 week, 8 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | -0.36 (0.09) | -0.36 (0.09) | -0.44 (0.09) | -0.63 (0.09)
  8-week change (n=28; n=37; n=39; n=37) | -2.43 (0.17) | -2.13 (0.15) | -2.23 (0.15) | -2.27 (0.15)

12. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at 1 Week and 8 Weeks
Description: The PGI-I Rating Scale was a 7-point scale: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; or 7=very much worse. Least squares (LS) Means were adjusted for treatment group, site, visit and treatment-by-visit interaction, gender, age, baseline score and baseline score-by-visit interaction and an unstructured covariance matrix.
Time Frame: 1 week, 8 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
units on a scale
  1-week change | 3.72 (0.13) | 3.77 (0.13) | 3.52 (0.13) | 3.47 (0.12)
  8-week change (n=28; n=37; n=39; n=37) | 2.31 (0.19) | 2.40 (0.17) | 2.36 (0.16) | 2.40 (0.16)

13. Secondary Outcome: Time to Onset of Nausea
Description: Events of nausea were taken from the adverse event (AE) data. Participants were censored based on the following rules: 1=study discontinuation date if the participant discontinues the study; 2=study lost to follow-up date if the participant drops out of the study.
Time Frame: Baseline to onset of nausea (Baseline up to 8 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 40 | 38 | 38 | 37
days | 2.0 [1.0 to 9.0] | 1.0 [1.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 7.0 [2.0 to 56.0] | 6.0 [1.0 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

14. Secondary Outcome: Time to Resolve Nausea
Description: as for outcome 13
Time Frame: Nausea onset up to nausea resolve (Baseline up to 8 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 33 | 25 | 27 | 30
days | 6.0 [4.0 to 9.0] | 8.0 [5.0 to 15.0] | 15.0 [9.0 to 22.0] | 6.0 [4.0 to 7.0]

15. Secondary Outcome: Percentage of Participants Achieving Response
Description: Response was defined as ≥50% decrease from baseline on the 17-item Hamilton Depression Rating Scale (HAMD-17) total score. HAMD-17 total scores ranged from 0 (not at all depressed)-52 (severely depressed).
Time Frame: Baseline up to 8 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
percentage of participants | 51.8 | 49.2 | 47.5 | 47.5

16. Secondary Outcome: Percentage of Patients Achieving Remission
Description: Remission was defined as 17-item Hamilton Depression Rating Scale (HAMD-17) total score ≤7. HAMD-17 total scores ranged from 0 (not at all depressed)-52 (severely depressed).
Time Frame: Baseline up to 8 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine 60 mg With Food | Duloxetine 60 mg Without Food | Duloxetine 30 mg With Food | Duloxetine 30 mg Without Food
Number analyzed (Participants) | 56 | 59 | 59 | 61
percentage of participants | 42.9 | 37.3 | 35.6 | 32.8

ADVERSE EVENTS:
Arm/Group | Duloxetine 30 mg With Food | Duloxetine 60 mg With Food | Duloxetine 30 mg Without Food | Duloxetine 60 mg Without Food
Serious Adverse Events (participants affected / at risk) | 1/63 | 1/59 | 2/64 | 0/63
Other Adverse Events (participants affected / at risk) | 52/63 | 55/59 | 57/64 | 58/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 30 mg With Food (N=63) | Duloxetine 60 mg With Food (N=59) | Duloxetine 30 mg Without Food (N=64) | Duloxetine 60 mg Without Food (N=63)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 30 mg With Food (N=63) | Duloxetine 60 mg With Food (N=59) | Duloxetine 30 mg Without Food (N=64) | Duloxetine 60 mg Without Food (N=63)
Palpitations (Cardiac disorders) | 0 (0) | 4 (4) | 2 (2) | 3 (3)
Vision blurred (Eye disorders) | 5 (5) | 1 (1) | 0 (0) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 6 (6) | 7 (7) | 4 (5)
Constipation (Gastrointestinal disorders) | 12 (12) | 9 (10) | 9 (10) | 10 (11)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (5) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 10 (11) | 10 (10) | 12 (12)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 4 (5) | 4 (4) | 2 (3)
Nausea (Gastrointestinal disorders) | 39 (42) | 41 (49) | 38 (43) | 39 (43)
Vomiting (Gastrointestinal disorders) | 2 (2) | 8 (8) | 8 (9) | 10 (10)
Asthenia (General disorders) | 4 (4) | 1 (1) | 5 (5) | 5 (6)
Decreased appetite (Metabolism and nutrition disorders) | 11 (12) | 11 (11) | 13 (13) | 11 (11)
Dizziness (Nervous system disorders) | 11 (11) | 8 (8) | 10 (10) | 7 (7)
Headache (Nervous system disorders) | 11 (11) | 10 (10) | 14 (16) | 8 (8)
Sedation (Nervous system disorders) | 5 (5) | 6 (6) | 5 (5) | 6 (6)
Somnolence (Nervous system disorders) | 0 (0) | 4 (4) | 5 (5) | 9 (10)
Tremor (Nervous system disorders) | 1 (1) | 4 (4) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 6 (7) | 4 (4) | 3 (3) | 6 (6)
Insomnia (Psychiatric disorders) | 8 (8) | 8 (9) | 6 (6) | 5 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 1 (1) | 5 (5)

LIMITATIONS AND CAVEATS:
Large number of protocol violations; bias due to unblinded, open-label design (participants were predisposed to expect an outcome of nausea as the primary endpoint); use of emetogenic medications; incorrect reporting and intake of food and drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days